CLINICAL TRIAL: NCT03956979
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study in Parkinson's Disease Patients With Moderate to Severe Dyskinesia to Assess the Efficacy and Safety/Tolerability of Two Dose Combinations of JM-010
Brief Title: A Study in Parkinson's Disease in Patients With Moderate to Severe Dyskinesia
Acronym: ASTORIA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Contera Pharma (Industry)
Collaborators: Bukwang Pharmaceutical (Industry)
Responsible Party: Sponsor
Organization: Bukwang Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JM-010CS03; 2017-003415-19 (EudraCT Number)
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Dyskinesias
MeSH Terms: conditions — Dyskinesias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, double-dummy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- JM-010 group A (Experimental): Group A (JM-010 dose fixed combination drug(tablet)) +Placebo 2
  Interventions: Drug: JM-010 group A
- JM-010 group B (Experimental): Group B (JM-010 8/0.8mg dose fixed combination drug(tablet)) + Placebo 1
  Interventions: Drug: JM-010 group B
- Placebo (Placebo Comparator): Double-dummy - 2 tablets = Placebo 1 +Placebo 2
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: JM-010 group A — JM-010 fixed combination drug (Group A) + Placebo 2
  Other Names: JM-010
  Arms: JM-010 group A
Drug: JM-010 group B — JM-010 fixed combination drug (Group B) + Placebo 1
  Other Names: JM-010
  Arms: JM-010 group B
Drug: Placebos — Placebo 1 + Placebo 2
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The current study will explore the efficacy, safety and tolerability of 2 dose combinations of JM-010 to determine the optimal doses of each component to be studied in confirmatory clinical trials.

DETAILED DESCRIPTION:
This is a Phase 2, double-blind, double-dummy, placebo-controlled, randomized, parallel group, multicentre study.

Subjects with a diagnosis of moderate to severe dyskinesia in Parkinson's disease (PD) will complete a Screening Visit to assess eligibility to participate in the study.

Subjects will continue with their usual levodopa treatment regimen for the duration of study participation.

The screening assessment period will be a minimum of 1 week up to a maximum of 6 weeks. Subjects deemed to be eligible at the end of the Screening Visit will be randomly assigned in a 1:1:1 ratio to receive either 1 of the 2 dose combinations of JM-010 and 1 placebo, or 2 placebos as per the double-dummy study design. The randomized subjects will be followed treatment periods for 12 weeks and safety follow periods for 2 weeks, including pharmacokinetic (PK) sub-study.

ELIGIBILITY:
Inclusion Criteria:

* Is able to read, understand, and provide written, dated informed consent prior to Screening Visit.
* Is male or female, between 18 and 80 years of age at Screening Visit.
* Is diagnosed with idiopathic PD that meets UK Parkinson's Disease Society (UKPDS) Brain Bank Clinical Diagnostic Criteria and requires treatment with and shows responsiveness to levodopa.
* Has experienced dyskinesia over a period of at least 3 months prior to Screening Visit
* Has stable peak-effect dyskinesia
* Has more than one hour of "ON" time with troublesome dyskinesia during daily waking hours on a 24-hour PD subject diary
* Is on a stable levodopa dosing regimen requiring at least 3 dose administrations but no more than 6 dose administrations per day

Exclusion Criteria:

* Has undergone surgery for the treatment of PD
* Has a current diagnosis of Substance Use (including alcohol) Disorder (Abuse or Dependence, as defined by Diagnostic and Statistical Manual, Fifth Edition [DSM 5]),
* Has psychiatric diagnosis of acute psychotic disorder or other psychiatric diagnoses
* Has a significant risk for suicidal behaviour in the opinion of the investigator during the course of their participation in the study
* Has current seizure disorders (other than febrile seizures in childhood) requiring treatment with anticonvulsants.
* Has known serious ongoing symptomatic cerebral disease or cerebrovascular disease or any acute brain trauma requiring treatment with anti-convulsant therapy within 5 years prior Visit 2, Week 0 (Baseline Visit).
* Has a history of exclusively diphasic, OFF state, myoclonic, dystonic, or akathetic dyskinesia without peak-dose dyskinesia.

Other criteria related to other medical conditions to be referred to the protocol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
Unified Dyskinesia Rating Scale (UDysRS) | 12 Weeks
  To compare the efficacy of JM-010 to that of placebo therapy in reducing dyskinesia severity in Parkinson's Disease by evaluating the total score mean change from Baseline to Week 12 in the sum of the items comprising UDysRS. The scoring range is 0-104, and a higher score indicates more severe dyskinesia.

SECONDARY OUTCOMES:
Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | 2 Weeks, 4 Weeks, 8 Weeks, 12 Weeks
  To compare the efficacy of JM-010 to that of placebo therapy as measured by the sum of the MDS-UPDRS Part III score changes from Baseline to Weeks 2, 4, 8, 12. The score range is 0-132, where a higher score means more severe motor impairment.
Clinician's Global Impression-Change (CGI-C) score | 12 Weeks
  To compare the efficacy of JM-010 to that of placebo therapy in relation to improvement in clinician-reported PD symptoms as measured by CGI-C score at Week 12. The CGI-C uses the following ratings: 0=not assessed; 1=very much improved; 2=much improved; 3=a little improved; 4=no change; 5=minimally worse; 6=much worse; and 7=very much worse.
Hauser diary | 2 Weeks, 4 Weeks, 8 Weeks, 12 Weeks
  To compare the efficacy of JM-010 to that of placebo therapy as measured by ON time without troublesome dyskinesia changes, OFF time changes, ON time with troublesome dyskinesia changes, Total time with dyskinesia changes from Baseline to Week 2, 4, 8, 12 in Hauser diary
Unified Dyskinesia Rating Scale (UDysRS) | 2 Weeks, 4 Weeks, 8 Weeks
  To compare the efficacy of JM-010 to that of placebo therapy in reducing dyskinesia severity in Parkinson's Disease by evaluating the total score mean change from Baseline to Week 2, 4, 8.
  The scoring range is 0-104, and a higher score indicates more severe dyskinesia.

CONTACTS AND LOCATIONS:
Overall Officials: Contera Clinical Development, Study Director — Contera Pharma
Locations (5):
- Contera Investigational site_FR, Toulouse, France
- Contera Investigational site_DE, Rostock, Germany
- Contera Investigational site_IT, Roma, Italy
- Contera Investigational site_KOR, Seoul, South Korea
- Contera Investigational site_ES, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McFarthing K, Prakash N, Simuni T. CLINICAL TRIAL HIGHLIGHTS - DYSKINESIA. J Parkinsons Dis. 2019;9(3):449-465. doi: 10.3233/JPD-199002. No abstract available. PMID 31356217